CLINICAL TRIAL: NCT02278497
Title: Assessment of Coronary Flow Reserve by PET-H215O and FFR in Patients Suspected of Coroanry Artery Disease. a Comparative Study With Dynamic Acquisition Using CZT Camera and 99mcTc-mibi.
Brief Title: Assessment of Coronary Flow Reserve by PET-H215O and FFR. Comparison With Dynamic Acquisition Using CZT Camera
Acronym: WATERDAY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Spectrum Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-006
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASSESSMENT OF CORONARY FLOW RESERVE BY PET-H215O AND FFR (Other)
  Interventions: Other: ASSESSMENT OF CORONARY FLOW RESERVE BY PET-H215O AND FFR

INTERVENTIONS:
Other: ASSESSMENT OF CORONARY FLOW RESERVE BY PET-H215O AND FFR

SUMMARY:
The study will assess coronary flow reserve by PET-H215O and FFR in patients suspected of coroanry artery disease. This a comparative study with dynamic acquisition using CZT camera and 99mcTc-mibi. 20 patients will have those measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 80 years
* Suspected coronary disease and / or coronary syndrome patient ST-
* Patient who has been informed of the study and has given his informed consent
* Patient affiliated to a social security system.

Exclusion Criteria:

* Patient having no coronary disease at coronary angiography with FFR on the 3 main epicardial arteries (absence of ≥ 50% stenosis of at least one artery)
* Delay of Care grater than 30 days between the PET and SPECT imaging and the diagnostic coronary angiography
* Patient with a recent history of myocardial infarction and STEMI, unstable angina
* Patient with extra-cardiac disease whose prognosis can interfere with the treatment decision
* Pregnant or lactating women
* Patient allergic to contrast products during coronary angiography
* Patient with MDRD clearance les than 60 ml / min
* Patient Under guardianship, or unable to understand the purpose of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Assess myocardial coronary reserve by cardiac CZT camera and Tcmibi comparing with the PET and the water marked during coronary FFR (Flow Fraction Reserve) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Medecine Nucleaire, Caen, France